CLINICAL TRIAL: NCT01144026
Title: Phase I/IIA Clinical Study of TUTI-16 in HIV-1 Infected and Uninfected Subjects
Brief Title: Clinical Study of TUTI-16 in HIV-1 Infected and Uninfected Subjects
Acronym: THYMON-10001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thymon, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THYMON-10001
Record Dates: First submitted 2010-06-12; First posted 2010-06-15 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infections
Keywords: HIV; vaccine; lipopeptide; Tat; TUTI-16; THYMON
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TUTI-16 (0.2mg) (Experimental): Two subcutaneous injections of 0.2 mg at Day 0, and Week 5.
  Interventions: Biological: TUTI-16 (0.2mg)
- TUTI-16 (1.0 mg) (Experimental): Two subcutaneous injections of 1.0 mg at Day 0, and Week 5.
  Interventions: Biological: TUTI-16 (1.0 mg)

INTERVENTIONS:
Biological: TUTI-16 (0.2mg) — Two subcutaneous injections of 0.2 mg at Day 0, and Week 5.
  Arms: TUTI-16 (0.2mg)
Biological: TUTI-16 (1.0 mg) — Two subcutaneous injections of 1.0 mg at Day 0, and Week 5.
  Arms: TUTI-16 (1.0 mg)

SUMMARY:
This protocol represents the second in human study of TUTI-16, and is being conducted to continue to gather safety and human immunogenicity (anti-HIV-1 Tat titers) data of subcutaneously administered TUTI-16.

DETAILED DESCRIPTION:
HIV-1 Tat protein, a virally encoded toxin, is secreted by HIV-1 infected cells and acts on uninfected cells, rendering them permissive for HIV-1 replication. HIV-1 Tat enhances chronic viral replication and induces immune suppression. Antibodies to Tat inhibit this Tat-mediated transcellular activation in vitro and minimize chronic plasma viremia. HIV-1 Tat activities can be blocked in vitro and in vivo by anti-Tat antibodies.

The Thymon Universal Tat Immunogen (TUTI-16) is a fully synthetic, self-adjuvanting lipopeptide vaccine that is water soluble and administered by subcutaneous injection. In preclinical studies, a priming dose and a three week boost in rats induced a high titer antibody response to the eight known distinct epitope variants of HIV-1 Tat protein. These antibodies block the function of the HIV-1 Tat protein (toxin), which is essential to the maintenance of chronic HIV-1 viremia. Therefore, TUTI-16 has potential as a therapeutic vaccine for HIV-1 in humans.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age ≥18 and ≤50 years at Screening
* HIV negative healthy subjects or HIV-1 seropositive subjects on effective ART for >2 months (undetectable HIV plasma viremia), viral set point before ART >3,000
* CD4+ T-cell count ≥ 500/mm3.

Exclusion Criteria:

* Pregnant/nursing females
* Positive for HBV or HCV
* Acute Herpetic event
* Any clinically significant out-of range laboratory value
* Routine or PRN consumption of immune suppressive medications that the subject is unable or unwilling to discontinue during the study
* Participation in another investigational drug/vaccine study within 30 days preceding the first injection of investigational agent in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardik Donikyan, MD, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs, New York, New York, United States

REFERENCES:
- [Derived] Goldstein G, Chicca JJ. Exploratory clinical studies of a synthetic HIV-1 Tat epitope vaccine in asymptomatic treatment-naive and antiretroviral-controlled HIV-1 infected subjects plus healthy uninfected subjects. Hum Vaccin Immunother. 2012 Apr;8(4):479-85. doi: 10.4161/hv.19184. Epub 2012 Feb 16. PMID 22336878

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TUTI-16 (0.2mg) | TUTI-16 (1.0 mg)
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TUTI-16 (0.2mg) | TUTI-16 (1.0 mg) | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.4 (8.51) | 36.4 (4.56) | 38.4 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Anti-Tat Antibody Titer
Description: ELISA based chemiluminescent assay to determine the anti-Tat antibody response
Time Frame: 5 weeks
Population: all participants enrolled were analyzed
Measure: Median (Full Range); unit: ng/mL
Arm/Group | TUTI-16 (0.2mg) | TUTI-16 (1.0 mg)
Number analyzed (Participants) | 10 | 5
ng/mL | 401 [0 to 2565] | 887 [99 to 2286]

ADVERSE EVENTS:
Arm/Group | TUTI-16 (0.2mg) | TUTI-16 (1.0 mg)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 4/10 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TUTI-16 (0.2mg) (N=10) | TUTI-16 (1.0 mg) (N=5)
injection site reaction (General disorders) | 4 (9) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No